CLINICAL TRIAL: NCT00397267
Title: Treatment of Acute Asthma in ER With Combination of Systemic Steroids and Inhaled Steroids
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOR440906CTIL
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2006-11-28 (Estimated); Status verified 2006-10

CONDITIONS: Asthma Exacerbation
Keywords: Dyspnea; Cough
MeSH Terms: conditions — Dyspnea; Cough

INTERVENTIONS:
Drug: inhalation of corticosteroids

SUMMARY:
We assume that the combination of systemic steroids and inhaled steroid in the first hour of treatment in the ER will decrease the admission rate and improve faster the pulmonary function.

120 patients refferd to the ER due to asthma attack aged 18-60 with PFR < 60% 0o predicted will participate in the study after giving informed consent.

The usual treatment in the ER is inhalation of Beta 2 short acting and I.V solumedrol 120 mg . The study group will recieve in addition 3 inhalation of Budesonide 1000 microgram each during the first hour.

The controlled group will recieve Nacl 0.9% PFR will be followed 0 30 60 120 min.

DETAILED DESCRIPTION:
Primary end points- PFT improvment and admission rate.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic patients aged 18-60 with PFR < 60% of predicted

Exclusion Criteria:

* Patients with other chronic diseases
* cardiac renal hepatic etc will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120
Dates: Start 2007-01; Study Completion 2007-12

PRIMARY OUTCOMES:
PFT improvment
Admission rate

CONTACTS AND LOCATIONS:
Overall Officials: Dov Heimer, M.D, Principal Investigator — BGU Soroka medical center
Locations (1):
- ER Soroka Med Center, Beersheba, Israel